CLINICAL TRIAL: NCT07075016
Title: Ivosidenib and Azacitidine With or Without Venetoclax in Adult Patients With Newly Diagnosed IDH1-Mutated AML or MDS/AML Considered Ineligible for Intensive Chemotherapy
Acronym: EVOLVE 1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Collaborators: German-Austrian Acute Myeloid Leukemia Study Group (Unknown); United Kingdom AML Research Network (Unknown); Gruppo Italiano Malattie EMatologiche dell'Adulto (GIMEMA) (Unknown); Swiss Group for Clinical Cancer Research (SAKK) (Unknown); Danish Acute Leukemia Group (Unknown); Grupo Cooperativo de Estudio y Tratamiento de las Leucemias Agudas y Mielodisplasias (Other); Nordic AML Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: HO173; 2024-512753-24 (EudraCT Number)
Record Dates: First submitted 2025-06-19; First posted 2025-07-20 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: IDH1; Newly AML diagnosed; Ineligible for intensive chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo comparator: Venetoclax-placebo (Placebo Comparator): day 1-28 Placebo Treatment will be on a continuous 28-day cycle schedule continued until disease relapse, disease progression, development of unacceptable toxicity, death, withdrawal of subject or other protocol defined criteria for discontinuation (which ever comes first)
  Interventions: Drug: Placebo
- Experimental: Venetoclax (Experimental): day 1-28 Venetoclax Treatment will be on a continuous 28-day cycle schedule continued until disease relapse, disease progression, development of unacceptable toxicity, death, withdrawal of subject or other protocol defined criteria for discontinuation (which ever comes first)
  Interventions: Drug: Venetoclax 400

INTERVENTIONS:
Drug: Venetoclax 400 — day 1-28 per cycle
  Arms: Experimental: Venetoclax
Drug: Placebo — day 1-28 per cycle
  Arms: Placebo comparator: Venetoclax-placebo

SUMMARY:
The standard treatment for patients with acute myeloid leukemia (AML) with an abnormality in the IDH1 gene, who are not eligible for intensive chemotherapy, is a combination of ivosidenib and azacitidine. In this study it is investigated whether adding venetoclax to the standard treatment can improve the outcome of the treatment of this specific form of AML. The safety is investigated and how well it works. In order to properly assess the value of venetoclax, the effect of venetoclax is compared with the effect of a placebo. A placebo is a product without an active ingredient, a 'fake medicinal product'.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with newly diagnosed IDH1-mutated AML, or IDH1-mutated MDS/AML according to the 2022 International Consensus Classification (Appendix A). Patients with AML with both IDH1 and IDH2 mutation are eligible as well. Of note: in case both NPM1 and IDH1 are mutated and both EVOLVE-1 (HO173/AMLSG 3423/ACT-HOV-AML-001) and EVOLVE-2 (HO177/AMLSG 35-24/ACT-HOV-AML-002are open for inclusion at your site, then patients can only be included in the EVOLVE-1 trial (HO173)
2. Central confirmation of IDH1 mutation in one of the dedicated central genetic laboratories.
3. Age ≥ 18 years, no upper age limit.
4. Patient is ineligible for intensive induction chemotherapy by meeting at least 1 of the following criteria:

   * older than or equal to 75 years of age ineligible for intensive chemotherapy per physician's discretion (with an ECOG performance status 0-2; Appendix C).
   * 18-74 years: patient is not eligible for standard chemotherapy because of any of the following co-morbidities: o ECOG performance status 2 or 3 (Appendix C). o Cardiac history of chronic heart failure requiring treatment; or with an ejection fraction ≤50%; or chronic stable angina.

     * DLCO ≤ 65% or FEV1 ≤ 65%.
     * Creatinine clearance ≥ 30 mL/min to <45 ml/min calculated by the Cockcroft Gault formula.
     * Moderate hepatic impairment with total bilirubin > 1.5 to < 3.0 x upper limit of normal (ULN).
     * Any other comorbidity that the local physician assesses to be incompatible with intensive chemotherapy. If a patient meets this criterion, sponsor must be informed via HO173@erasmusmc.nl
5. Patient must have a projected life expectancy of at least 12 weeks (as assessed by the treating physician).
6. Patient must have a white cell blood (WBC) count of < 25 x 109/L. Hydroxyurea can be used prior to study enrollment to reduce the WBC count to meet this criterion.
7. Adequate renal function as evidenced by serum creatinine ≤ 2.0 × upper limit of normal (ULN) or creatinine clearance >30 mL/min based on the Cockcroft-Gault glomerular filtration rate (GFR).
8. Adequate hepatic function as evidenced by:

   * Serum total bilirubin ≤ 3.0 × ULN unless considered due to Gilbert's disease, or leukemic involvement. If a patient meets this criterion, sponsor must be informed via HO173@erasmusmc.nl Page 30 of 117 HOVON 173 AML / AMLSG 34-23 / ACT-HOV-AML-001 Version 1.1, UK 11 FEB 2025
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 3.0 × ULN, unless considered due to leukemic involvement. If a patient meets this criterion, sponsor must be informed via HO173@erasmusmc.nl
9. Female patients :

   * of nonchildbearing potential must be: o postmenopausal (defined as at least 1 year without any menses). o documented surgically sterile (e.g. documented hysterectomy, bilateral oophorectomy or bilateral salpingectomy) or status posthysterectomy (at least 1 month prior to screening).
   * of childbearing potential (not surgically sterile and not postmenopausal) must agree to avoid pregnancy during the study and for 6 months after the final study drug administration o and have a negative urine or serum pregnancy test at screening.

     o and, if heterosexually active, agree to consistently apply one highly effective* method of birth control in combination to a barrier method for the duration of the study and for 6 months after the final study drug administration.
   * must agree not to breastfeed starting at screening and throughout the study period, and for 1 month after the final study drug administration.
   * must agree not to donate ova starting at screening and throughout the study period, and for 6 months after the final study drug administration.
10. Men must use a latex condom during any sexual contact with women of childbearing potential (WOCBP), even if they have undergone a successful vasectomy and must agree to avoid to father a child (while on therapy and for 6 months after the final study drug administration). In addition, their female partners of childbearing potential must use a highly effective method of birth control.
11. Male patient must not donate sperm starting at screening and throughout the study period and for 6 months after the final study drug administration.
12. Able to understand and willing to sign an informed consent form (ICF).
13. Institutional Review Board/Independent Ethics Committee-approved written informed consent and privacy language as per national regulations must be obtained from the participant prior to any study-related procedures (including consent for withdrawal of prohibited medication, if applicable).

Exclusion Criteria:

1. Subject has previously been treated for AML; a treatment period with hydroxyurea to control WBC counts is allowed; prior treatment with a hypomethylating agent for MDS-EB is not allowed; prior treatment with erythropoiesis-stimulating agents or luspatercept for MDS is allowed.
2. Acute promyelocytic leukemia (APL) with t(15;17)(q24.1;q21.2); PML-RARA; or one of the other pathognomonic variant chromosomal translocations / fusion genes.
3. AML with BCR-ABL1; or myeloid blast crisis of CML
4. Significant active cardiac disease within 3 months prior to the start of study treatment, including:

   - New York Heart Association (NYHA) class III or IV congestive heart failure (Appendix F)

   - Myocardial infarction

   - Unstable angina
   * Severe cardiac arrhythmias
   * Congenital long QT syndrome of family member with this condition
   * QTcF >480 msec on screening electrogram (mean of triplicate recordings).
5. Familial history of sudden death or polymorphic ventricular arrhythmia.
6. Severe obstructive or restrictive ventilation disorder.
7. History of stroke or intracranial hemorrhage within 6 months prior to randomization.
8. Clinical symptoms suggestive of active central nervous system (CNS) leukemia or known CNS leukemia. Evaluation of cerebrospinal fluid (CSF) during screening is only required if there is a clinical suspicion of CNS involvement by leukemia during screening.
9. Active infection, including hepatitis B or hepatitis C or Human Immunodeficiency Virus (HIV) infection, that is uncontrolled prior to first dose of study treatment and may interfere with the study objectives or which could expose the patient to undue risk through the participation in the clinical trial; an infection controlled with an approved antibiotic/ antiviral/ antifungal treatment that is not a strong or moderate CYP3A inducer is allowed. Patients with COVID-19 infection can be enrolled, if the patient has no symptoms and was tested negative twice by PCR test prior to inclusion in the trial.
10. Immediate life-threatening, severe complications of leukemia such as uncontrolled bleeding and/or disseminated intravascular coagulation.
11. Conditions that limit the ingestion or gastrointestinal absorption of orally administered drugs
12. Patient with a currently active second malignancy. Patients are not considered to have a currently active malignancy, if they have completed therapy and are considered by their physician to be at < 30% risk of relapse within one year. However, patients with the following history/concurrent conditions are allowed:

    * Basal or squamous cell carcinoma of the skin;
    * Carcinoma in situ of the cervix;
    * Carcinoma in situ of the breast;
    * Incidental histologic finding of prostate cancer.
13. Receipt of live, attenuated vaccine within 30 days prior to the study inclusion (NOTE: patient, if enrolled, should not receive live vaccine during the study and until 6 months after the therapy).
14. Severe neurological or psychiatric disorder interfering with ability to give an informed consent.
15. Contraindication to any of the anti-leukemic agents used (as per SmPC). 16. Participation in other prospective studies with anti-leukemic and/or investigational agents.

17. Patient taking Dabigatran unless they can be transferred to other medications within ≥5 half-lives prior to dosing. Patients taking other P-gP transporter-sensitive medications (see Appendix J) should be properly monitored during the study if they cannot be transferred to other medications." 18. Patients taking known strong cytochrome P450 (CYP) 3A4 inducers (see Appendix H), unless they can be transferred to other medications within ≥5 half-lives prior to dosing.

19. The patient is a pregnant or lactating woman, or plans to become pregnant during the study.

20. Patient who has once been screened and randomized into this HO173 trial but was considered ineligible cannot re-enter this trial at a later date.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) in patients with newly diagnosed IDH1-mutated AML ineligible for intensive chemotherapy | 12 months after inclusion of last AML patient
  Event-free survival (EFS) in patients with newly diagnosed IDH1-mutated AML ineligible for intensive chemotherapy, measured from the date of randomization to the date of treatment failure, hematologic relapse from CR/CRh or death from any cause, whichever occurs first. Treatment failure is defined as lack of obtaining either CR or CRh by week 24. Patients evaluable for response but not achieving CR or CRh by week 24 will be considered a treatment failure at day 1 post randomization to avoid ambiguities of variable or prolonged periods without response. Patients who die before week 24 without response assessments will also be considered treatment failures at day 1 post randomization. Patients who are alive but not evaluable for response will be censored at day 1 post randomization. Patients who achieved CR or CRh by week 24 and are not known to have morphologic relapse or died will be censored at the date of the last clinical assessment.

SECONDARY OUTCOMES:
Overall survival (OS) in patients with newly diagnosed IDH1-mutated AML | 12 months after inclusion of last AML patient
  Overall survival (OS) in patients with newly diagnosed IDH1-mutated AML, measured from the day of randomization to the date of death from any cause; patients not known to have died are censored on the date they were last known to be alive.
Rate of CR/CRh in patients with newly diagnosed IDH1-mutated AML | 12 months after inclusion of last AML patient
  Rate of CR/CRh in patients with newly diagnosed IDH1-mutated AML, defined as the proportion of patients with CR/CRh at any time point during protocol therapy.
Rate of CR in patients with newly diagnosed IDH1-mutated AML | 12 months after inclusion of last AML patient
  Rate of CR in patients with newly diagnosed IDH1-mutated AML, defined as the proportion of patients with CR at any time point during protocol therapy.
Rate of CR/CRi in patients with newly diagnosed IDH1-mutated AML | 12 months after inclusion of last AML patient
  Rate of CR/CRi in patients with newly diagnosed IDH1-mutated AML, defined as the proportion of patients with CR/CRi at any time point during protocol therapy.
Rates of CR, CR/CRh and CR/CRi without measurable residual disease as assessed by multicolor flow cytometry | 12 months after inclusion of last AML patient
  Rates of CR, CR/CRh and CR/CRi without measurable residual disease as assessed by multicolor flow cytometry (CRMRD-, CR/CRhMRD- and CR/CRiMRD-) in patients with newly diagnosed IDH1-mutated AML, defined as the proportion patients with CRMRD-, CR/CRhMRD- and CR/CRiMRD-, respectively, at any time point during protocol therapy.
Time to achievement of response (CR, CR/CRh and CR/CRi) in patients with newly diagnosed IDH1-mutated AML | 12 months after inclusion of last AML patient
  Time to achievement of response (CR, CR/CRh and CR/CRi) in patients with newly diagnosed IDH1-mutated AML, defined as time from the date of randomization until the 1st occurrence of response.
Duration of response (CR, CR/CRh and CR/CRi) in patients with newly diagnosed IDH1mutated AML | 12 months after inclusion of last AML patient
  Duration of response (CR, CR/CRh and CR/CRi) in patients with newly diagnosed IDH1mutated AML, measured from the date of achievement of a response until the date of hematologic relapse or death from any cause; patients without any of these events will be censored on the date of last clinical assessment.
The rate of transfusion independence (platelets and RBC) in patients with newly diagnosed IDH1-mutated AML | A period of at least 56 days with no transfusion between the first dose of study drug and the last dose of study drug + 30 days.
  The rate of transfusion independence (platelets and RBC) in patients with newly diagnosed IDH1-mutated AML, defined as the proportion of patients who achieved transfusion independence; transfusion independence is defined as a period of at least 56 days with no transfusion between the first dose of study drug and the last dose of study drug + 30 days.

CONTACTS AND LOCATIONS:
Locations (119):
- Austria (3):
  - AT-Feldkirch-IKHF, Feldkirch
  - AT-Salzburg-SALK, Salzburg
  - AT-Vienna-HANUSCH, Vienna
- Belgium (8):
  - BE-Antwerpen-ZAS, Antwerp
  - BE-Brussel-BORDET, Brussels
  - BE-Brussel-UZBRUSSEL, Brussels
  - BE-Bruxelles-STLUC, Brussels
  - BE-Gent-UZGENT, Ghent
  - BE-Leuven-UZLEUVEN, Leuven
  - BE-Liege-CHULIEGE, Liège
  - BE-Yvoir-MONTGODINNE, Yvoir
- Denmark (5):
  - DK-Aalborg-AALBORGUH, Aalborg
  - DK-Aarhus N-AUH, Aarhus N
  - DK-Copenhagen-RIGSHOSPITALET, Copenhagen
  - DK-Odense-OUH, Odense
  - DK-Roskilde-ROSKILDE, Roskilde
- Estonia (2):
  - EE-Tallinn-REGIONAALHAIGLA, Tallinn
  - EE-Tartu-TARTU, Tartu
- Finland (2):
  - FI-Helsinki-HUS, Helsinki
  - FI-Tampere-TAYS, Tampere
- France (14):
  - FR-Angers-CHUANGERS, Angers
  - FR-Pessac Cedex-CHUBORDEAUX, Bordeaux
  - FR-Caen-CHUCAEN, Caen
  - FR-Créteil cedex-CHUMONDOR, Créteil
  - FR-Grenoble cedex 9-CHUGRENOBLE, Grenoble
  - FR-Lille-CHULILLE, Lille
  - FR-Lyon Pierre Benite cedex-LYONSUD, Lyon
  - FR-Montpellier-CHUSAINTELOIS, Montpellier
  - FR-Nantes-CHUNANTES, Nantes
  - FR-Nice-LARCHET, Nice
  - FR-Rennes cedex 9-CHURENNES, Rennes
  - FR-Rouen cedex-BECQUEREL, Rouen
  - FR-Saint-Priest-en-Jarez-STETIENNE, Saint-Etienne
  - FR-Le Chesnay cedex-CHVERSAILLES, Versailles
- Germany (26):
  - DE-Berlin-CAMPUSBENFRANKLIN, Berlin
  - DE-Berlin-CAMPUSVIRCHOW, Berlin
  - DE-Berlin-VIVANTESNEUKOLLN, Berlin
  - DE-Bochum-RUB, Bochum
  - DE-Bonn-UNIBONN, Bonn
  - DE-Braunschweig-KLINIKUMBRAUNSCHWEIG, Braunschweig
  - DE-Bremen-KBM, Bremen
  - DE-Darmstadt-KLINIKUMDARMSTADT, Darmstadt
  - DE-Flensburg-MALTESER, Flensburg
  - DE-Freiburg-UNIKLINIKFREIBURG, Freiburg im Breisgau
  - DE-Greifswald-UNIGREIFSWALD, Greifswald
  - DE-Halle-UMH, Halle
  - DE-Hamburg-ASKLEPIOSSTGEORG, Hamburg
  - DE-Hamburg-UKE, Hamburg
  - DE-Hannover-MHHANNOVER, Hanover
  - DE-Hannover-SILOAHKRH, Hanover
  - DE-Heilbronn-SLK, Heilbronn
  - DE-Karlsruhe-KLINIKUMKARLSRUHE, Karlsruhe
  - DE-Mainz-UNIMEDIZINMAINZ, Mainz
  - DE-Minden-MUEHLENKREISKLINKEN, Minden
  - DE-München-IRZTUM, München
  - DE-Oldenburg-KLINIKUMOLDENBURG, Oldenburg
  - DE-Regensburg-UKR, Regensburg
  - DE-Stuttgart-KLINIKUMSTUTTGART, Stuttgart
  - DE-Tübingen-MEDUNITUEBINGEN, Tübingen
  - DE-Ulm-UNIKLINKULM, Ulm
- Ireland (4):
  - IE-Cork-CUH, Cork
  - IE-Dublin 7-MATER, Dublin
  - IE-Dublin 8-ST JAMES, Dublin
  - IE-Galway-UHGALWAY, Galway
- Italy (5):
  - IT-Bologna-MALPHIGI, Bologna
  - IT-Milano-NIGUARDA, Milan
  - IT-Roma-SAPIENZA, Roma
  - IT-Roma-TORVERGATA, Roma
  - IT-Torino-CITTADELLASALUTE, Torino
- LT-Vilnius-SANTA, Vilnius, Lithuania
- Netherlands (14):
  - NL-Den Bosch-JBZ, 's-Hertogenbosch
  - NL-Amsterdam-VUMC, Amsterdam
  - NL-Arnhem-RIJNSTATE, Arnhem
  - NL-Breda-AMPHIA, Breda
  - NL-Dordrecht-ASZ, Dordrecht
  - NL-Eindhoven-CATHARINA, Eindhoven
  - NL-Enschede-MST, Enschede
  - NL-Sittard-Geleen-ZUYDERLAND, Geleen
  - NL-Groningen-UMCG, Groningen
  - NL-Nijmegen-RADBOUDUMC, Nijmegen
  - NL-Rotterdam-ERASMUSMC, Rotterdam
  - NL-DenHaag-HAGA, The Hague
  - NL-Utrecht-UMCU, Utrecht
  - NL-Zwolle-ISALA, Zwolle
- Norway (4):
  - NO-Bergen-HELSEBERGEN, Bergen
  - NO-Oslo-OSLOUH, Oslo
  - NO-Tromsø-NORTHNOORWEGEN, Tromsø
  - NO-Trondheim-STOLAV, Trondheim
- Spain (5):
  - ES-Barcelona-CLINICUB, Barcelona
  - ES-Barcelona-GERMANTRIALS, Barcelona
  - ES-Barcelona-SANTPAU, Barcelona
  - ES-Girona-ICSTRUETA, Girona
  - ES-Valencia-MALVARROSA, Valencia
- Sweden (4):
  - SE-Goteborg-SAHLGRENSKA, Gothenburg
  - SE-Lund-SUH, Lund
  - SE-Stockholm-KAROLINSKAHUDDINGE, Stockholm
  - SE-Uppsala-UPPSALAUH, Uppsala
- Switzerland (4):
  - CH-Basel-USB, Basel
  - CH-Bellinzona-IOSI, Bellinzona
  - CH-Bern-INSEL, Bern
  - CH-Zurich-USZ, Zurich
- United Kingdom (18):
  - UK-Birmingham-QE, Birmingham
  - UK-Blackpool-BLACKPOOLVICTORIA, Blackpool
  - UK-Bristol-BRISTOLCENTRE, Bristol
  - UK-Cardiff-UHW, Cardiff
  - UK-Glasgow-BEATSON, Glasgow
  - UK-Leeds-STJAMESUH, Leeds
  - UK-Leicester-LEICESTERRI, Leicester
  - UK-London-KCH, London
  - UK-London-ROYALMARSDEN, London
  - UK-London-UNICOLLEGEHOSP, London
  - UK-Manchester-CHRISTIE, Manchester
  - UK-Manchester-ROYALINFIRMARY, Manchester
  - UK-Newcastle on Tyne-FREEMAN, Newcastle upon Tyne
  - UK-Nottingham-NOTTINGHAMCH, Nottingham
  - UK-Oxford-CHURCHILL, Oxford
  - UK-Portsmouth-QUEENALEXANDRA, Portsmouth
  - UK-Southampton-SOUTHAMPTONGH, Southampton
  - UK-Wolverhampton-NEWCROSSH, Wolverhampton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: HOVON website — https://www.hovon.org